CLINICAL TRIAL: NCT04595760
Title: Factors Influencing Fertility or Pregnancy Health
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000058; 000058-E
Record Dates: First submitted 2020-10-20; First posted 2020-10-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-02

CONDITIONS: Menstrual Cycles; Conception; Early Pregnancy Loss; Pregnancy Outcomes
Keywords: Pregnancy; Fertility; Reproductive Health; Fecundability; Natural History
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EPS Study Participants: Women who participated in the 1982-1986 North Carolina Early Pregnancy Study (EPS)

SUMMARY:
Background:

The North Carolina Early Pregnancy Study (EPS) was held from 1982 to 1986. Women who were trying to get pregnant took part in the study. They collected urine samples. They kept diaries. They filled out surveys. They answered questions about their partners. They were asked about their drug use. Data about air pollution and other exposures were also collected. A follow-up study was held from 2010 to 2011. Researchers want to use the data and samples to study factors that affect reproductive success.

Objective:

To examine behavioral and environmental exposures and reproductive health, such as menstrual cycles, conception, pregnancy loss, and pregnancy outcomes.

Eligibility:

The 221 healthy women age 21-42 who were planning to get pregnant and took part in the 1982-86 North Carolina EPS at the time they stopped using all birth control. A 2010-11 follow-up included 173 of these women.

Design:

This study uses existing data. No new data will be collected in this study.

Stored urine samples may be used. Data from surveys and other sources will be used. All of the women who gave data and samples will be included.

Electronic data is held in secure databases. The data is kept on computers that are password protected. Hard-copy data are stored in locked file cabinets.

The study will take place at more than one site. Data will be shared with groups outside the NIH....

DETAILED DESCRIPTION:
Existing self-reported data and assay results from the 1982-1986 North Carolina Early Pregnancy Study (EPS) and a subsequent 2010-2011 cohort follow-up study will be used to examine predictors of fertility and pregnancy outcomes. Some of these data will be harmonized with data from other studies by our collaborator (Harville PI, Tulane University) to examine factors, such as marijuana use in women and their partners, influencing reproductive success, including (but not limited to) conception, pregnancy loss, and birth outcomes. Women enrolled in the original EPS study after discontinuing birth control and were followed for the occurrence of a pregnancy. Participants completed daily diaries and collected first morning urine specimens which allowed the identification of hormonal endpoints. Thus, each woman s time to pregnancy was prospectively measured. In the EPS Follow-up study, women completed a questionnaire that included their recall of their time to pregnancy during the study. This allowed analysis of two major questions, one regarding the recall of time- to-pregnancy, and the other regarding the natural length of gestation. Several exposure metrics based on address geolocation data were calculated, including the distance from residence to nearest major road, air pollution and related exposures, light at night, and other exposures. Existing urine specimens can be assayed for numerous environmental contaminants including metals, pesticides, and drug metabolites (both over-the-counter medications like acetaminophen and drugs of abuse like marijuana or opioids). Urine specimens can also be used to examine nutritional markers such as phytoestrogen exposure and caffeine metabolites. Additional hormone measures may also be possible as metabolomics and technology improve. Thus, the stored EPS specimens can be leveraged to answer multiple, relevant fertility research questions. Women in the original tudy answered questions regarding their tobacco smoking and marijuana smoking. In addition, partners of the women were asked the same series of questions regarding tobacco and marijuana use.

We intend to use all of this existing data, assay results, and to perform additional urine assays, to examine factors influencing reproductive success, including (but not limited to) conception, pregnancy loss, and birth outcomes. To address some of these questions, de-identified data from the Early Pregnancy Study will be harmonized with data from other studies in the Preconception Period Analysis of Risks and Exposures Influencing Health and Development (PrePARED) consortium. Further, de-identified data and specimens will be shared with Dr. Ashley Boggs and colleagues to address the objectives below. Data and specimens will be shared with other qualified investigators in the future to address relevant research questions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* healthy white women aged 21-42 who were planning to become

pregnant

-women enrolled in the 1982-1986 North Carolina Early Pregnancy

Study (EPS) at the time they discontinued all methods of birth control

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who participated in the 1982-1986 North Carolina Early Pregnancy Study (EPS)
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Time-to-pregnancy | Prospectively measured
  Reproductive function includes a spectrum of relevant endpoints and outcomes. We will examine behavioral and environmental exposures and reproductive health including menstrual cycles, conception, pregnancy loss, and pregnancy outcomes

SECONDARY OUTCOMES:
Pregnancy loss, hormone levels, birth outcomes, pregnancy complications | Prospectively measured
  Reproductive function includes a spectrum of relevant endpoints and outcomes. We will examine behavioral and environmental exposures and reproductive health including menstrual cycles, conception, pregnancy loss, and pregnancy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Z Jukic, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institute of Environmental Health Sciences (NIEHS), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided